CLINICAL TRIAL: NCT00864422
Title: Driving Plasticity in the Motor Brain in Chronic Back Pain
Brief Title: Changes in Motor Cortex Following Exercises for Chronic Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Dr Henry Tsao, Centre for Clinical Research Excellence in Spinal Pain, Injury and Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NHMRC-ID351656; NHMRC-ID401599; PRF-007/06
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; motor training; motor cortex; brain plasticity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Skilled motor training
- 2 (Active Comparator)
  Interventions: Behavioral: Walking exercise

INTERVENTIONS:
Behavioral: Skilled motor training — This involves training subjects to independently and cognitively activate the deep abdominal muscles, transversus abdominis, with minimal or no activity in other trunk muscles. The contraction is held for 10 seconds and subjects complete three blocks of ten contractions, twice per day for two weeks. This training protocol is commonly used clinically for people with chronic back pain.
  Arms: 1
Behavioral: Walking exercise — The control intervention involves walking exercises for ten minutes, twice per day. Subjects are advised to walk at their own pace with no instructions on activation of specific trunk muscles. The exercise is performed over two weeks.
  Arms: 2

SUMMARY:
The motor cortex of the brain changes following chronic pain and injury, and this is linked to pain-associated changes in motor behaviour. This study aimed to investigate whether therapeutic exercises in patients with chronic pain can induce reorganisation of the motor cortex and restore normal motor behaviour. The investigators hypothesised that motor training can induce reorganisation of the motor cortex and that these changes are related to improved motor behaviour.

DETAILED DESCRIPTION:
The sensory and motor systems can reorganize following injury and learning of new motor skills. Recently we observed adaptive changes in motor cortical organization in patients with chronic back pain, which are closely linked to changes in motor behavior. Although pain-related alterations in behavior can be trained and are associated with improved symptoms, it remains unclear whether these meaningful functional outcomes are related to motor cortical reorganization. Here we investigate the effects of two interventions in people with chronic back pain: skilled motor training and a control intervention of self-paced walking exercise. We measured motor cortical excitability (motor threshold (MT)) and organization (center of gravity (CoG) and map volume) of the deep abdominal muscle, transversus abdominis (TrA), using transcranial magnetic stimulation (TMS). In addition, motor behavior of TrA was assessed during single rapid arm movements. The study helps to elucidate the mechanisms of specific motor exercises in chronic back pain management.

ELIGIBILITY:
Inclusion Criteria:

* Sustained or episodic non-specific low back pain lasting longer than 3 months

Exclusion Criteria:

* Orthopaedic, neurological, circulatory or respiratory conditions
* History or family history of epilepsy
* Recent or current pregnancies
* Previous surgery to the abdomen or back
* Abdominal or back exercises in the preceding 12 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Motor cortical map and excitability from transcranial magnetic stimulation | Pre and 2 weeks post-intervention

SECONDARY OUTCOMES:
Motor activation of the abdominal muscles during functional arm movement task | Pre and 2 weeks post-intervention
Self-reported pain (VAS scale) and functional scale (patient-specific functional scale) | Pre and 2 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Hodges, MedDr (Neurosci) PhD BPhty, Study Director — The University of Queensland; Henry Tsao, PhD MPhty (Manipulative) BPhty, Principal Investigator — The University of Queensland
Locations (1):
- Centre for Clinical Research Excellence in Spinal Pain, Injury and Health, Brisbane, Queensland, Australia